CLINICAL TRIAL: NCT00937729
Title: Prospective Evaluation Among Patients Infected by HIV 1 in Virological Failure Owing to Lack of Compliance, of the Benefit in Terms of Compliance of an Optimised Antiretroviral Treatment Containing Enfuvirtide (Fuzeon) Associated With Two Active Molecules
Brief Title: Prospective Evaluation Among Patients Infected by HIV 1 in Virological Failure Owing to Lack of Compliance, of the Benefit in Terms of Compliance of an Optimised Antiretroviral Treatment With Enfuvirtide (Fuzeon) Associated With Two Active Molecules
Acronym: AMPHORE
Status: Terminated | Type: Observational
Why Stopped: difficult to include patients
Sponsor: University Hospital, Rouen (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: 2008/122/HP
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Last update posted 2012-02-16 (Estimated); Status verified 2012-02

CONDITIONS: HIV1 Infection; HIV Infections
Keywords: uncompliant patients with virological failure; Treatment experienced
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- enfuvirtide: all patients would received enfuvirtide and and optimised background

SUMMARY:
In case of lack of compliance in HIV1 patients, the investigators hope to prove that enfuvirtide injection during almost 3 months, with nurse help at home and therapeutic education may contribute to obtain a good compliance more than 95% in these patients.

ELIGIBILITY:
Inclusion Criteria:

* virological failure, more than 18 years, prouved lack of compliance, with no sub-optimal treatment, in ambulatory status.

Exclusion Criteria:

* hospitalization,HIV2 infection,pregnancy,preliminary treatment with enfuvirtide,chimiotherapy , opportunistic infection in progress

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients HIV1 infected in virological failure (viral load > 50 copies/ml) by lack of compliance,old of more than 18 years, who never received enfuvirted and without opportunistic infection, yet treated by almost one molecule of each group.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2009-06; Primary Completion 2011-01 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
viral load compliance | one year

SECONDARY OUTCOMES:
statistical analysis of MOS HIV | one year

CONTACTS AND LOCATIONS:
Overall Officials: BORSA-LEBAS Françoise, Principal Investigator — CHU Hôpitaux de Rouen
Locations (1):
- Borsa-Lebas, Rouen, France